CLINICAL TRIAL: NCT05530954
Title: Clinical Evaluation of Direct Pulp Capping in Primary Molars
Brief Title: Direct Pulp Capping in Primary Molars
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nayera tarek, PhD researcher of Pediatric Dentistry and Dental Public Health, Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DPC in primary molars
Record Dates: First submitted 2022-09-03; First posted 2022-09-07 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Direct Pulp Capping
Keywords: primary dentition; MTA; Dycal; bioactive material; deciduous dentition; Direct pulp capping
MeSH Terms: interventions — mineral trioxide aggregate; MTA Bio; Dycal

STUDY DESIGN:
Intervention Model Description: After informed consent, baseline clinical and radiographic assessment will be obtained and recorded in patient examination sheet. Participants who met the inclusion criteria were randomly allocated to two groups (n = 26/group, N = 52 in total) according to the capping martials using the envelope randomization method. All patients were recalled and their treated molars were evaluated clinically and radiographically at 3months, 6months, 9months ,12months follow up periods.
  2 study groups according to capping material that will be used (Dycal or MTA) and each group will be divided to 2 subgroups according to site of exposure axial or pulpal
Who Masked: Participant
Masking Description: capping material used
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mineral trioxide aggregate (MTA) (Active Comparator): * where the pulp tissue is exposed during final caries removal, hemostasis will be achieved by cavity irrigation with sterile saline solution for up to 4 minutes till control of bleeding
  * Teeth with pulp exposure less than 1mm in diameter surrounded by sound dentin will be candidates for direct pulp capping
  * Following the removal of the saline, the exposed pulp will be irrigated with 17% EDTA solution (Prevest Direct, India) for 1 minute
  * According to site of exposure, the groups will be further subdivided into Group A (n=13) with exposure in pulpal floor and Group B (n=13) with exposure in axial wall of the cavity.
  * Exposed pulp will be covered with fast set MTA paste after cavity dryness with sterile cotton pellet then the tooth will be restored with Self-cured glass ionomer restorative material (SDI Riva self-cure, Australia) and tooth will be covered by stainless steel crown
  Interventions: Other: Mineral trioxide aggregate (MTA)
- Hard setting Calcium Hydroxide (Dycal) (Active Comparator): * where the pulp tissue is exposed during final caries removal, hemostasis will be achieved by cavity irrigation with sterile saline solution for up to 4 minutes till control of bleeding
  * Teeth with pulp exposure less than 1mm in diameter surrounded by sound dentin will be candidates for direct pulp capping
  * Following the removal of the saline, the exposed pulp will be irrigated with 17% EDTA solution (Prevest Direct, India) for 1 minute
  * According to site of exposure, the groups will be further subdivided into Group A (n=13) with exposure in pulpal floor and Group B (n=13) with exposure in axial wall of the cavity.
  * Exposed pulp will be covered with Dycal paste after cavity dryness with sterile cotton pellet then the tooth will be restored with Self-cured glass ionomer restorative material (SDI Riva self-cure, Australia) and tooth will be covered by stainless steel crown
  Interventions: Other: Hard setting Calcium Hydroxide (Dycal)

INTERVENTIONS:
Other: Mineral trioxide aggregate (MTA) — Materials for Vital Pulp Capping
  Other Names: BIO MTA; CERKAMED, Poland
  Arms: Mineral trioxide aggregate (MTA)
Other: Hard setting Calcium Hydroxide (Dycal) — Materials for Vital Pulp Capping
  Other Names: Dycal; Promedica Urbical, Germany
  Arms: Hard setting Calcium Hydroxide (Dycal)

SUMMARY:
The purpose of this study is to Assess the effect of MTA and hard setting Calcium Hydroxide (Dycal) on the clinical and radiographic outcome of direct pulp capping in primary molars and evaluate overall success rate of direct pulp capping in primary molars.

DETAILED DESCRIPTION:
After informed consent, baseline clinical and radiographic assessment will be obtained and recorded in patient examination sheet.

Participants who met the inclusion criteria were randomly allocated to two groups (n = 26/group, N = 52 in total) according to the capping martials using the envelope randomization method.

2 study groups according to capping material that will be used (Dycal or MTA) and each group will be divided to 2 subgroups according to site of exposure axial or pulpal.

All patients were recalled and their treated molars were evaluated clinically and radiographically at 3months, 6months, 9months ,12months follow up periods.

ELIGIBILITY:
Inclusion Criteria:

* Cooperative child and compliant parent.
* Complete physical and mental health.
* Children who are known to be healthy and free from systemic diseases.
* Primary molars with deep carious lesions leading to pathological exposure but with no signs or symptoms of irreversible pulpitis or necrosis such as spontaneous pain, tenderness to percussion, abscess, fistula, periodontal tissue swelling, or abnormal tooth mobility.

Exclusion Criteria:

* A deep carious lesion in close proximity to the pulp with an intact lamina dura.
* Absence of widening of periodontal membrane space or radiolucency at the furcation and periapical region.
* Absence of pulpal calcifications, obliteration of the pulp and root canal, or internal/external root resorption.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-27 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
clinical success of direct pulp capping treatment after 3 months follow up | 3 months
  Presence of any of these clinical findings will be considered failure:
  pain on mastication or spontaneous pain, as reported by the patient, without clinical evidence of plaque retention around the crown margin denoting bad oral hygiene.
  pain on percussion on clinical examination . non-physiologic mobility. fistula or sinus tract.
clinical success of direct pulp capping treatment after 6 months follow up | 6 months follow up
  Presence of any of these clinical findings will be considered failure:
  pain on mastication or spontaneous pain, as reported by the patient, without clinical evidence of plaque retention around the crown margin denoting bad oral hygiene.
  pain on percussion on clinical examination . non-physiologic mobility. fistula or sinus tract.
clinical success of direct pulp capping treatment after 9 months follow up | 9 months follow up
  Presence of any of these clinical findings will be considered failure:
  pain on mastication or spontaneous pain, as reported by the patient, without clinical evidence of plaque retention around the crown margin denoting bad oral hygiene.
  pain on percussion on clinical examination . non-physiologic mobility. fistula or sinus tract.
clinical success of direct pulp capping treatment after 12 months follow up | 12 months follow up
  Presence of any of these clinical findings will be considered failure:
  pain on mastication or spontaneous pain, as reported by the patient, without clinical evidence of plaque retention around the crown margin denoting bad oral hygiene.
  pain on percussion on clinical examination . non-physiologic mobility. fistula or sinus tract.
radiographic success of direct pulp capping treatment after 3 months follow up | 3 months follow up
  the absence of the following radiographic findings indicate the success of capping material in pulp therapy:
  * pathological internal or external root resorption.
  * PDL widening.
  * inter-radicular radiolucency formation postoperatively.
  * periapical radiolucency formation postoperatively.
radiographic success of direct pulp capping treatment after 6 months follow up | 6 months follow up
  the absence of the following radiographic findings indicate the success of capping material in pulp therapy:
  * pathological internal or external root resorption.
  * PDL widening.
  * inter-radicular radiolucency formation postoperatively.
  * periapical radiolucency formation postoperatively.
radiographic success of direct pulp capping treatment after 9 months follow up | 9 months follow up
  the absence of the following radiographic findings indicate the success of capping material in pulp therapy:
  * pathological internal or external root resorption.
  * PDL widening.
  * inter-radicular radiolucency formation postoperatively.
  * periapical radiolucency formation postoperatively.
radiographic success of direct pulp capping treatment after 12 months follow up | 12 months follow up
  the absence of the following radiographic findings indicate the success of capping material in pulp therapy:
  * pathological internal or external root resorption.
  * PDL widening.
  * inter-radicular radiolucency formation postoperatively.
  * periapical radiolucency formation postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: S M Awad, PhD/Prof, Study Chair — Head of Pediatric Dentistry and Dental Public Health, Mansoura University; A Y El Hosainy, PhD, Study Director — Lecturer of Pediatric Dentistry, Faculty of Dentistry, Mansoura University; N T El Saied, MSc, Principal Investigator — PhD researcher at Faculty of Dentistry, Mansoura University
Locations (1):
- Outpatient clinic of the Department of Pediatric Dentistry, Faculty of Dentistry- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Caicedo R, Abbott PV, Alongi DJ, Alarcon MY. Clinical, radiographic and histological analysis of the effects of mineral trioxide aggregate used in direct pulp capping and pulpotomies of primary teeth. Aust Dent J. 2006 Dec;51(4):297-305. doi: 10.1111/j.1834-7819.2006.tb00447.x. PMID 17256303
- [Result] Faraco IM Jr, Holland R. Response of the pulp of dogs to capping with mineral trioxide aggregate or a calcium hydroxide cement. Dent Traumatol. 2001 Aug;17(4):163-6. doi: 10.1034/j.1600-9657.2001.170405.x. PMID 11585142
- [Result] de Lourdes Rodrigues Accorinte M, Reis A, Dourado Loguercio A, Cavalcanti de Araujo V, Muench A. Influence of rubber dam isolation on human pulp responses after capping with calcium hydroxide and an adhesive system. Quintessence Int. 2006 Mar;37(3):205-12. PMID 16536148
- See also: © European Academy of Paediatric Dentistry 2018 — http://doi.org/10.1007/s40368-018-0360-x